CLINICAL TRIAL: NCT03643536
Title: Effects of a 12-week Exercise-based Program on Quality of Life in Myocardial Revascularization Subjects With Normal and Reduced Left Ventricular Ejection Fraction
Brief Title: 12-week Exercise-based Program in Myocardial Revascularization Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación del Caribe para la Investigación Biomédica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018200801
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2014-01

CONDITIONS: Quality of Life
Keywords: left ventricular ejection fraction; quality of life

STUDY DESIGN:
Intervention Model Description: A prospective controlled before-after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-WPEP in subjects with reduce LVEF (Experimental): Intervention: a 12 week physical exercise program in the health-related quality of life of CABG or PCI subjects with LVEF by 2D-echocardiography between 30-54%. The quality of life was measured using SF-36 questionnaire
  Interventions: Other: 12-WPEP
- 12-WPEP in subjects with normal LVEF (Active Comparator): Intervention: a 12 week physical exercise program in the health-related quality of life of or PCI subjects with LVEF by 2D-echocardiography≥ 55% (control group)The quality of life was measured using SF-36 questionnaire
  Interventions: Other: 12-WPEP

INTERVENTIONS:
Other: 12-WPEP — The 12-WPEP (week physical exercise program) was carried out in 3 sessions each 40 or 60minutes with alternate days per week during 3 months, and with an intensity between 40 to 80 percent of their VO2 max, as the AHA recommends

SUMMARY:
To determine if a 12-week physical exercise program (12-WPEP), after percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) with different left ventricular ejection fraction (LVEF) might improve the health-related quality of life (HRQOL).

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) and coronary artery bypass graft surgery (CABG) are interventions that can reduce cardiovascular symptoms such as dyspnea and angina. The life quality and the functional capacity improved in the subjects who underwent surgery. However, new cardiac events, death and obstruction of the bypass placed can exist. To diminish these risks, national and international guides recommend cardiac rehabilitation (CR) for people with coronary disease, who have suffered a myocardial infarction and are subjected to CABG and PCI. A 20-30% reduction of morbidity and mortality can be obtained with the use of CR. According to the European Society of Cardiology (ESC), the American Heart Association (AHA) and the American College of Cardiology (ACC), CR is a recommendation Class Type I, in subjects treated with PCI and CABG. This includes prescribed physical exercises, education, and counseling to modify the effects of coronary heart disease and improve long-term survival. Exercise-based cardiac rehabilitation is an effective and safe therapy to be used in the management of clinically stable patients following PCI or CABG. The maximum oxygen uptake (VO2max) is improved by the exercise carried out during CR, optimizing the physical condition and health-related quality of life (HRQOL).

The HRQOL is considered a very important criterion used to evaluate the effectiveness of different treatments in patients with coronary disease, and is defined by subjective evaluation regarding the current activities of health care and health promotion; it indicates the personal perception in various aspects such as the recovery of the functional, labor, sexual and social capabilities of the patient, factors that have great importance in the evolution of the patient; this perception is considered the best indicator of quality of life, and has become a key concept for the decision making. In this study, we will evaluate the effects of a physical exercise program in the health-related quality of life of subjects following CABG or PCI with normal and reduced left ventricular ejection fraction (LVEF)

ELIGIBILITY:
Inclusion Criteria:

- CABG or post-PCI subjects and agreed to participate by signing the informed consent form.

Exclusion Criteria:

* Subjects with musculoskeletal limitations for physical exercise, untreated ventricular arrhythmias, with the presence of residual pericardial effusion, history of intermittent claudication or left ventricular ejection fraction <30% measured by 2D-echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01-01; Primary Completion 2014-12-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQOL) | 12 weeks after the inclusion
  For the evaluation of health-related quality of life, 36 health survey questionnaire (SF-36) was used. This questionnaire has 36 questions that address two major components based on 8 fields: physical component which includes physical functioning, physical performance, pain and general health, and the mental component which includes vitality, social function, emotional role and mental health.To calculate the score, the items for each one of the eight dimensions are encoded, added and transformed into a scale from 0 (worst health status for this dimension) to 100 (best health status).

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Urina-Triana, PhD ( c), Study Director — Fundacion del Caribe para la Investigacion Biomedica; Mirary Mantilla-Morron, Principal Investigator — Fundacion del Caribe para la Investigacion Biomedica
Locations (1):
- Fundacion del Caribe para la Investigacion Biomedica (Fundacion Bios), Barranquilla, Atlántico, Colombia